CLINICAL TRIAL: NCT06526338
Title: A Randomized Phase 2 Study to Evaluate the Safety and Efficacy of IP-001 as Adjuvant Therapy in Participants With Hepatocellular Carcinoma After Complete Radiological Response After Surgical Resection and Local Ablation or Local Ablation Alone
Brief Title: Adjuvant IP-001 Treatment for HCC Patients Following Surgical Resection and Ablation or Ablation Alone
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Robert C. Martin (Other)
Responsible Party: Sponsor-Investigator, Robert C. Martin, Director of the Division of Surgical Oncology Robert C. Martin, University of Louisville
Organization: University of Louisville (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24.0321
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — N-dihydrogalactochitosan; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IP-001 (Experimental): 1.0% IP-001 for injection immediately following local ablation or surgical resection and local ablation
  Interventions: Drug: 1.0% IP-001 for injection; Procedure: Surgical Resection and Local Ablation; Procedure: Local Ablation Alone
- Control (Active Comparator): Local ablation or surgical resection and local ablation alone
  Interventions: Procedure: Surgical Resection and Local Ablation; Procedure: Local Ablation Alone

INTERVENTIONS:
Drug: 1.0% IP-001 for injection — Participants will receive a single injection of 1.0% IP-001 following local ablation or surgical resection and local ablation
  Arms: IP-001
Procedure: Surgical Resection and Local Ablation — Participants will undergo surgical resection of the tumor and local ablation by either radiofrequency ablation (RFA ) or microwave ablation (MWA)
Procedure: Local Ablation Alone — Participants will have local ablation of the tumor by either radiofrequency ablation (RFA) or microwave ablation (MWA) alone

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a single injection of IP-001 as adjuvant therapy after local ablation or surgical resection and ablation in patients with hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
This is a Phase 2, two-armed, randomized study designed to evaluate the safety and efficacy of a single administration of intratumoral IP-001 injection following local ablation or surgical resection and local ablation in patients with hepatocellular carcinoma who have an intermediate or high risk of recurrence compared to curative ablation or ablation and surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of signing Informed Consent.
* Has a diagnosis of hepatocellular carcinoma (HCC) documented radiologically by American Association for the Study of Liver Diseases (AASLD) criteria and/or histopathologically from a tumor biopsy.
* Has a treatment plan to receive either a curative ablation (RFA or MWA) or a curative surgical resection and ablation.
* Has HCC with intermediate, high or very high risk of recurrence.
* Has hepatic only HCC (disease confined to the liver only), defined by no extra-hepatic lesions greater than 1 cm in size.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Patient with past or ongoing hepatitis C virus (HCV) infection will be eligible if the patient has completed HCV treatment at least 1 month prior to Day 1.
* Patient with controlled hepatitis B will be eligible if the patients meets the following criteria:

  1. Antiviral therapy for hepatitis B virus (HBV) must be given for at least 4 weeks and HBV viral load must be less than 500 IU/mL prior to treatment. Patients on active HBV therapy with viral loads under 00 IU/mL should stay on the same therapy throughout study treatment.
  2. Patients who are hepatitis B core antibody (anti-HBc) positive, negative for HBsAg, and negative or positive for anti- HBs, and who have an HBV viral load under 500 IU/mL do not require HBV anti-viral prophylaxis.
* Has adequate organ function as specified in the Adequate Organ Function Laboratory Values Table. Specimens must be collected within 14 days prior to Day 1.

Exclusion Criteria:

* Known allergic reaction to shellfish, crabs, crustacean, or any trial components.
* Has an active infection requiring systemic therapy.
* Has a diagnosis of immunodeficiency or currently receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent), or any other form of immunosuppressive therapy within 7 days prior to treatment day (Day 1), or has plans to start treatment including >10 mg daily of prednisone equivalent or any immunotherapy.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents or immunosuppressive drugs). NOTE: replacement therapy (e.g., thyroxine or insulin) is not considered a form of systemic treatment and is allowed.
* Has had an allogenic tissue/solid organ transplant.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, active tuberculosis, or idiopathic pneumonitis.
* Has received local therapy to liver, ablation other than radiofrequency or microwave ablation (i.e., alcohol ablation, transcatheter chemoembolization, transcatheter embolization, hepatic arterial infusion, local radiation/Stereotactic Body Radiation Therapy or radioembolization) less than 3 months prior to treatment.
* Is receiving any of the following prohibited concomitant therapies less than 21 days from treatment or 5 drug elimination half-lives, whichever is shorter prior to randomization:

  1. Antineoplastic systemic chemotherapy or biological therapy.
  2. Immunotherapy not specified in this protocol.
  3. Systemic glucocorticoids for any purpose other than to modulate symptoms from an adverse event (AE) that is suspected to have an immunologic etiology. Inhaled or topical steroids are allowed, and systemic steroids at doses ≤10 mg/day prednisone or equivalent are allowed. Exception: steroids may be used for premedication prior to imaging.
* Has received a live vaccine within 28 days prior to treatment Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival | From Date of Randomization until date of documented progression, assessed up to 60 months
  Radiological assessments (Triphasic CT or MRI) of the chest, abdomen and pelvis will occur every 12 weeks for the first 2 years, then every 24 weeks thereafter. Recurrence will be determined by the investigator's radiological review per RECIST v1.1

SECONDARY OUTCOMES:
Cancer Free Survival | Months 12 and 24
  Participants will be followed every 12 weeks from treatment Day 1 for the first 2 years, and every 24 weeks thereafter until disease related death.
Overall Survival | Months 12 and 24
  Participants will be followed every 12 weeks from treatment Day 1 for the first 2 years, and every 24 weeks thereafter until death of any cause.
Overall Survival Rate | Months 12 and 24
  Proportion of participants who have not experienced death from treatment Day 1 at 12 and 24 months after treatment.
Recurrence Free Survival Rate | Months 12 and 24
  Assessed from treatment Day 1 to documentation of disease recurrence or extrahepatic) or death, whichever occurs first.
Time to Intrahepatic Tumor Recurrence | From Date of Randomization until date of documented progression, assessed up to 60 months
  Radiological assessments (Triphasic CT or MRI) of the chest, abdomen and pelvis will occur every 12 weeks for the first 2 years, then every 24 weeks thereafter. Recurrence will be determined by the investigator's radiological review per RECIST v1.1
Time to Extrahepatic Tumor Recurrence | From Date of Randomization until date of documented progression, assessed up to 60 months
  Radiological assessments (Triphasic CT or MRI) of the chest, abdomen and pelvis will occur every 12 weeks for the first 2 years, then every 24 weeks thereafter. Recurrence will be determined by the investigator's radiological review per RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Robert CG Martin, MD, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No